CLINICAL TRIAL: NCT04517487
Title: Vaginal Microbiome Transplantation for Recurrent Bacterial Vaginosis-A Placebo, Randomized, Controlled Trial
Brief Title: Vaginal Microbiome Transplantation for Recurrent Bacterial Vaginosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Principal Investigator, Ahinoam Lev-Sagie, Principal investigator, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMO-19-691
Record Dates: First submitted 2020-08-15; First posted 2020-08-18 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Bacterial Vaginoses
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VMT recipients (Active Comparator): In order to prevent transfer of pathogens, sperm, or antibiotic-resistant commensals we will establish a "vaginal fluid bank" in which samples from suitable donors will be kept for future use:
  * Donors will be screened using a questionnaire addressing risk factors for potentially transmissible infections, undergo screening for cervico-vaginal infections, cervical cytology screening, and serology analysis for transmittable infections {see detailed screening in Lev-Sagie et al. Nat Med. 2019;25(10):1500-1504. doi: 10.1038/s41591-019-0600-6.}
  * The collected samples for VMT will be examined for bacteria,viruses and sperm.
  Before transplantation, patients will be treated with intravaginal antibiotics. A frozen specimen will be thawed at room temperature and will be placed in the patient's vagina.
  Following VMT, patients will be evaluated every 14 days for the first 2 months, then every month for additional 10 months.
  Interventions: Biological: Vaginal Microbiome Transplantation (VMT)
- Placebo (Placebo Comparator): Vaginal fluid of all recipients will be collected before initiation of the study using the same protocol, will be clearly labeled and will be kept frozen in similar conditions. These samples will be used in the placebo arm for autologous vaginal fluid transplantation.
  Before transplantation, patients will be treated with intravaginal antibiotic.
  Following Placebo, patients will be evaluated every 14 days for the first 2 months, then every month for additional 2-4 months.
  After 4-6 months, patients who initially received placebo will be offered a VMT in case they are still symptomatic and fulfill inclusion criteria, in an open-label phase.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Vaginal Microbiome Transplantation (VMT) — Healthy donors vaginal fluid is introduced into recipients' vagina to replace their indigenous disease-associated microbiome
  Arms: VMT recipients
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Vaginal Microbiome Transplantation (VMT) may be beneficial in treating the most severe cases of recurrent and antibiotics-nonresponsive cases of BV. Recently, we completed a preliminary study in which we treated patients with recurrent and antibiotics-non-responsive, intractable BV, with VMT from healthy donors [Lev-Sagie, Nature Medicine 2019]. Four VMT recipients in this preliminary study featured a significant improvement of both clinical symptoms and dysbiotic vaginal microbiome composition and function, which persisted over a long follow-up period, while one recipient featured a partial remission.

The proposed study is designed as a placebo, randomized controlled trial, and is aimed to further assess whether VMT may serve as a viable option in symptomatic, intractable BV. In the suggested study, we plan to compare transplantation of: 1) vaginal fluid from healthy donors, and 2) autologous transplantation, of the patient's own vaginal fluid.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50
* Recurrent BV, defined as ≥4 symptomatic episodes of BV during the last year, who require maintenance antibiotic treatment (twice weekly) in order to remain symptom-free, or if they experienced recurrence of BV in ≤ 2 months following antibiotic treatment, with a documented history of recurrent BV in the last year.
* Patients are otherwise healthy.
* Contraception use

Exclusion Criteria:

* Pregnancy or a planned pregnancy in the upcoming year
* Infection with HIV.
* Immunodeficiency status.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical parameters- patient's complains | 12 months
  Number of participants reporting disappearance of discharge and odor
Laboratory parameters- Amsel criteria | 12 months
  Presence or absence of each Amsel criteria (discharge, pH>4.5, positive whiff test and clue cells on microscopy)/
Vaginal fluid microscopy | 12 months
  Presence of Lactobacillus-dominant microbiome on microscopy
Microbiome composition | 12 months
  Characterization of the vaginal microbial community using shotgun analysis and16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Ahinoam Lev-Sagie, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lev-Sagie A, Goldman-Wohl D, Cohen Y, Dori-Bachash M, Leshem A, Mor U, Strahilevitz J, Moses AE, Shapiro H, Yagel S, Elinav E. Vaginal microbiome transplantation in women with intractable bacterial vaginosis. Nat Med. 2019 Oct;25(10):1500-1504. doi: 10.1038/s41591-019-0600-6. Epub 2019 Oct 7. PMID 31591599